CLINICAL TRIAL: NCT02733172
Title: Profiling Vulvodynia Based on Neurobiological and Behavioral Endophenotypes
Acronym: Vulvodynia
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jennifer Labus, PhD, PhD, University of California, Los Angeles
Other Study IDs: 13-001113
Record Dates: First submitted 2015-12-02; First posted 2016-04-11 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Vulvodynia
Keywords: Vulvodynia; Endophenotypes; functional MRI
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators plan to extensively phenotype a large sample of Vulvodynia (VD) patients using functional and structural brain imaging together with genetic, physiological, and biological parameters.

DETAILED DESCRIPTION:
Vulvodynia (VD) is a chronic pain disorder affecting up to 15% of women and resulting in substantial impairment in health-related quality-of-life. The treatment of the disorder is hampered by a lack of knowledge regarding its neurobiological basis. The proposed study is based on the general hypothesis that like other persistent pain conditions, VD clinical phenotypes (characteristic of the disorder) are composed of multiple biological endophenotypes (such as an hereditary characteristic that is normally associated with a condition but not a direct symptom of that condition) and that meaningful subgroups can be identified.

In the current proposal, the investigators plan to extensively phenotype a large sample of VD patients using functional and structural brain imaging together with genetic, physiological, and biological parameters. The hypothesis is that central mechanisms (including alterations in the processing/modulation of interoceptive signals from the external genitals) are important determinants of the clinical presentation, and that differences in these brain signatures could play an important role in treatment responsiveness. Such phenotyping has considerable implications for future drug development.

There will be a total of 100 females diagnosed with either generalized vulvodynia (GVD) or provoked vestibulodynia (PVD) which is similar however more localized to just the vestibule area of the vulva enrolled. It will be a total of 140 with PVD and 60 with GVD.

The study will involve 2 visits total over about 1-3 weeks depending on schedules and menstrual cycle. The investigators will not scan a person if menstruating AND having abdominal cramps/emotional liability as this may confound analysis.

The participant will be screened for inclusion /exclusion criteria. After signing the consent the participant will have a history and physical and brief psychological interview to evaluation for any psychological problems present (using standard DSM-IV (diagnostic and statistical manual for mental disorders) criteria. The participant will completed questionnaires to assess mood, pain, pain related behavior and sexual functioning on Survey Monkey. The participant will have a neuro-sensory evaluation of the perineum performed by a qualified gynecologist Medical Doctor or Nurse Practitioner. During the examination the clinician will swab the vaginal canal using 2 sterile swabs (vaginal fluid) for microbiota (normal vaginal healthy bacteria). There will be 1 venous blood draw of about 2 teaspoons via venipuncture by the nurse, to look at blood metabolites and genes. Then the participant will have discomfort threshold testing of the right and left shin and upper arm muscle with an algometer.

Following screening the participant will return within 1-3 weeks to have brain scanning done which involves both functional (resting state) and structural scans. The investigators will measure changes in the autonomic nervous system simultaneously through electrodes on finger tips which measure minute changes in sweat glands. Saliva samples will be collected for analysis of polymorphism in genes controlling inflammation, pain, and nerve functioning. Prior to the scanning the participant will be asked to complete questionnaires to assess current (state) mood and symptoms on Survey Monkey.

The length of time of each visit is assessed to be about 90 minutes each.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Female (VD is a disorder that affects women only).
2. Age: 18 to 55 years of age.
3. Language: Participants must be fluent in English, as demonstrated by verbal skills sufficient to participate in a conversation, including the ability to ask and answer questions at a level that assures adequate understanding of the study.
4. History of VD: Participants will be required to meet criteria for VD based on history and examination: At least 3 month history of pain, burning, or irritation, with an intensity of 4/10 or greater of the vulva either localized to the vestibule and precipitated by contact of the vestibule (Provoked VD) or located in other regions of the vulva (called GVD). The pain must not be attributable to dermatitis, dermatosis, candida, hormonal changes, or vaginitis.
5. Generally healthy without current neurological, cardiovascular, hepatic, renal, autoimmune diseases, diabetes or cancer.
6. Willingness to use acceptable contraceptive methods (e.g., hormonal, barrier, or sterilization) if sexually active.
7. Limited tobacco use allowed as described: must smoke less than 1/3 packs per day (5-6 cigarettes/day allowed) and also to be able to abstain from smoking for no less than 12 hours before MRI without any concern for nicotine craving.

Exclusion Criteria:

1. Psychiatric disease: Psychiatric criteria (DSM-IV) will be used to determine exclusion of volunteers with psychiatric illnesses. A psychological interview by a trained clinician to determine diagnoses. We will exclude participants with any disorders or psychiatric diagnoses, including, but not limited to; schizophrenia, bipolar disorder, current/active and untreated depression or generalized anxiety, post traumatic stress disorder, attention deficit hyperactive disorder, past history of eating disorders without successful treatment within 3 yrs, will not be allowed.
2. History of Drug Abuse (including major nicotine dependence): We will also exclude volunteers who give self- reports or other evidence of recent (within 6 months) use of psychotropic agents (other than light marijuana or alcohol). Meeting diagnostic criteria for current abuse or dependence on alcohol or any illicit drugs of abuse will be exclusionary.
3. Heavy tobacco smokers will be excluded to avoid confounding effects of nicotine withdrawal or recent smoking on assessments during functional MRI.
4. Medications or treatments for VD, including psychological or physical therapy, that have been initiated less than 3 months prior to the study. Topical medication such as gabapentin or estrogens are allowed. Limited use of certain antidepressants (tricyclics and serotonin inhibitors) will be allowed.
5. CNS disease: Evidence of central nervous system (CNS), cerebrovascular, and/or infectious disease, and history of neurological disease (e.g., stroke/epilepsy) or history of head trauma with loss of consciousness >30 minutes, any history of post-traumatic amnesia, or more than one episode of head trauma, regardless of severity.
6. Claustrophobia: Subjects will be questioned about their potential discomfort with enclosed spaces, such as an MRI scanner.

   Subjects reporting problems with enclosed spaces will be excluded.
7. Pregnancy: subjects will be required to have a pregnancy test on the day of the MRI scan.
8. Presence in the body of a metal device (e.g., pacemaker, infusion pump, aneurysm clip, metal prosthesis or plate) that could either interfere with the acquisition of the MRI scan of the brain or for whom the MRI scan would pose a potential risk will be excluded.
9. Postmenopausal women defined as no menses for 12 consecutive months.
10. Past medical history of other chronic pain disorders such as Irritable bowel syndrome, frequent migraines (weekly) or fibromyalgia; UNLESS vulvodynia is clearly the main pain disorder. The PI will determine if eligible.
11. Oral opiates/anxiolytics and steroids are never allowed due to changes in the brain that would confound analysis.
12. Morbid Obesity (BMI > 35%)
13. Current use of certain oral contraceptives, nuvaring, Intrauterine devices (IUD) or spermicide as contraceptive method.
14. Use of antibiotics, antifungal or probiotics within 6 weeks of study enrollment.
15. Engaging in vaginal penetration (such as sexual intercourse, douches, tampons) or use of fragranced feminine hygiene products within 7 days of study enrollment.
16. Recent or active bacterial or fungal infections within 6 weeks of study enrollment.
17. Menstrual cycle beginning within 1 week of study participation.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women 18-55 yo with vestibulodynia, and or generalized vulvodynia, characterized by at least 3 months history of pain, burning, or irritation, with an intensity of 4/10 or greater, of the vulva localized to the vestibule (vestibulodynia) with or without pain located in outer region of the vulva (generalized VD).
  The pain must NOT be attributable to current bacterial, fungal, or yeast infections, a skin condition (eg; dermatitis), hormonal changes, or vaginitis.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-07; Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Brain morphometry measured by magnetic resonance imaging (MRI) | Length of the brain imaging scans is 35 minutes; assessed 1 time
  Structural MRI collected to quantify these measures
Functional connectivity measured by magnetic resonance imaging (MRI) | Length of the brain imaging scans is 35 minutes; assessed 1 time
  Functional MRI collected to quantify these measures

SECONDARY OUTCOMES:
Genotyping for candidate gene polymorphism | 5 minutes at screening for saliva sample collecteion
  Genotyping for candidate gene polymorphism related to hypothalamic-pituitary-adrenal (HPA) axis function.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Labus, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Oughourlian TC, Tun G, Antony KM, Gupta A, Mays VM, Mayer EA, Rapkin AJ, Labus JS. Symptom-associated alterations in functional connectivity in primary and secondary provoked vestibulodynia. Pain. 2023 Mar 1;164(3):653-665. doi: 10.1097/j.pain.0000000000002754. Epub 2022 Aug 15. PMID 35972459